CLINICAL TRIAL: NCT06396364
Title: Third Generation Cryotherapy Reduces Time to Surgery and Local Complication in Patients With Ankle Fractures: a Prospective Randomized Controlled Trial
Brief Title: Cryotherapy Reduces Time to Surgery and Local Complication in Patients With Ankle Fractures
Acronym: Cryotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera San Camillo Forlanini (Other)
Responsible Party: Principal Investigator, Alessio Giai Via, M.D., Orthopaedic Sugeon, principal investigator, Azienda Ospedaliera San Camillo Forlanini
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: cryotherapy012021.n01
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Ankle Fractures
Keywords: cryotherapy; ankle fracture; ankle surgery; time to surgery; surgical site infections
MeSH Terms: conditions — Ankle Fractures; Surgical Wound Infection | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Patients were randomized in two groups at the time of the diagnosis in the emergency department. The treatment group (T: 89 patients) were treated with a third-generation cryotherapy device (Z- One®, Zamar) which was applied daily for 2 hours two times a day up to the day of surgery. The leg was immobilized in a walking boot which was removed when the cryotherapy device was applied. The control group (C: 80 patients) did not use cryotherapy before surgery, the leg was immobilized into a half cats and elevation of the injured limb was indicated.
  Pain was evaluated according to the Visual Analogue Scale (VAS) and the analgesic drug demand (including morphine or acetaminophen). The Bod
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy (Experimental): Patients were treated with a third-generation cryotherapy device (Z- One®, Zamar) which was applied daily for 2 hours two times a day up to the day of surgery. The leg was immobilized in a walking boot which was removed when the cryotherapy device was applied.
  Interventions: Device: Cryotherapy
- Immobilization and elevation (Active Comparator): The leg was immobilized into a half cats and elevation of the injured limb was indicated before surgery.
  Interventions: Device: Cryotherapy

INTERVENTIONS:
Device: Cryotherapy — Treatment group: the ankle was immobilized in a walking boot, then a third-generation cryotherapy device (Z- One®, Zamar) was applied daily for 2 hours two times a day up to the day of surgery. The walking boot was removed when the cryotherapy device was applied.
  Other Names: Third generation cryotherapy

SUMMARY:
Ankle fractures are common injuries and cryotherapy is routinely used to reduce pain, swelling and local skin complications, both before and after surgery. However, the results on ankle surgery are contradictory. Despite the benefits of cryotherapy in the pre- and postoperative care of ankle surgery, lack of standardized protocols and few level-1 studies make difficult to appreciate the effectiveness. In addition, there's scarce evidence on the benefits from the preoperative use of cryotherapy.

The aim of this study is to report the results with the use of third generation cryotherapy in the preoperative treatment of ankle fractures. Third generation devices use computed cryotherapy to deliver gradual changes in pressure and temperature. The software produces a progressive drop in temperature and a controlled slow return to room temperature environment, avoiding reactive vasodilation. Time to surgery, pain, opioids intake, and local skin complications have been investigated.

Methods 169 patients with ankle fracture were randomized in two groups, the cryotherapy group (89 patients) and the control group (C: 80 patients). The time-to- surgery, Visual Analogue Scale (VAS) and the analgesic drug demand (including morphine or acetaminophen) were recorded. The development of skin complications was assessed daily. BMI and number of cigarettes smoked were also recorded.

DETAILED DESCRIPTION:
The aim of this study is to assess the effects of third generation cryotherapy on time to surgery, pain, opioids intake, and local skin complications. Although the use of cryotherapy is traditionally believed to reduce pain, swelling, local skin complications and the need of analgesia, the results on ankle surgery are not well reported and still contradictory. The working hypothesis is that third generation cryotherapy is a safe, reduces time to surgery and is useful in the surgical management of ankle fractures The investigators analyzed the prospectively collected data of 169 patients with ankle fracture, treated with open reduction and internal fixation (ORIF). Patients were randomized in two groups at the time of the diagnosis in the emergency department. The treatment group (T: 89 patients) were treated with a third-generation cryotherapy device (Z- One®, Zamar) which was applied daily for 2 hours two times a day up to the day of surgery. The leg was immobilized in a walking boot which was removed when the cryotherapy device was applied. The control group (C: 80 patients) did not use cryotherapy before surgery, the leg was immobilized into a half cats and elevation of the injured limb was indicated. Patients were collected in two different hospitals (Azienda Ospedaliera San Camillo Forlanini -Roma and Ospedale San Paolo - Civitavecchia) between 2021 and 2023. All patients had signed a written consent, and the study was approved by the local ethic committee.

After the diagnosis was made and surgical treatment was indicated, the patient was hospitalized in the department of orthopedic and trauma surgery.

A power analysis was performed to evaluate the sample size necessary to guarantee a power of at least 0.9 with a significance level of 0.05 using preliminary data on time to surgery.

Univariate descriptive analysis of the variables under study was carried out by calculating the centrality and variability indices for the quantitative variables and frequency tables for the variables.

The homogeneity of the control group and the treatment group for the variables sex, age, type of fracture, diabetes, hypercholesterolemia, venous insufficiency, and BMI class were checked. Depending on the nature of the variables, a t-test or a chi-square test was used.

Any significant differences between the treatment and control groups were assessed using independent samples t-tests for quantitative variables and chi-square tests for qualitative variables. Where the sample size was not sufficient, the non-parametric Mann-Whitney test for independent samples was used.

An alpha significance level of 0.05 was used in all analyses mentioned. For the statistical analysis of data, IBM SPSS Statistics software version 28 was used

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency department with an ankle fracture

Exclusion Criteria:

* Open fractures
* Fracture-dislocations which required external fixation
* Patients with one or more associated fractures
* Patients with a diagnose of major trauma
* Patients who were not able to complain with the pre- and post-surgical indications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
time to surgery | From enrollment to surgery
  hours

SECONDARY OUTCOMES:
VAS Score | 6 hours
  VAS Score - Visual analogue scale. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 (pain as bad as it it could possibly be).
Skin complications | up to surgery
  The onset of preoperative skin complication as skin blisters have been recorded. complications
Morphine intake | up to surgery
  Pain was evaluated as the number of Morphine vials intake

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Pipino, M.D., Prof., Study Chair — San Raffaele University, Milan
Locations (2):
- Italy (2):
  - A.O. San Camillo Forlanini, Rome
  - A.O. San camillo Forlanini, Rome

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: the will be available with the published manuscript, or by asking to the corresponding author under reasonable request with no time restriction
Access Criteria: contacting the corresponding author (Alessio Giai Via) by e-mail
URL: https://crioterapiaortopedica.it/z-one/

REFERENCES:
- [Result] Herrera E, Sandoval MC, Camargo DM, Salvini TF. Motor and sensory nerve conduction are affected differently by ice pack, ice massage, and cold water immersion. Phys Ther. 2010 Apr;90(4):581-91. doi: 10.2522/ptj.20090131. Epub 2010 Feb 25. PMID 20185615
- [Result] Helmerhorst GT, Lindenhovius AL, Vrahas M, Ring D, Kloen P. Satisfaction with pain relief after operative treatment of an ankle fracture. Injury. 2012 Nov;43(11):1958-61. doi: 10.1016/j.injury.2012.08.018. Epub 2012 Aug 16. PMID 22901424
- [Result] Wilke B, Weiner RD. Postoperative cryotherapy: risks versus benefits of continuous-flow cryotherapy units. Clin Podiatr Med Surg. 2003 Apr;20(2):307-22. doi: 10.1016/S0891-8422(03)00009-0. PMID 12776983
- [Result] Douzi W, Guillot X, Bon D, Seguin F, Boildieu N, Wendling D, Tordi N, Dupuy O, Dugue B. 1H-NMR-Based Analysis for Exploring Knee Synovial Fluid Metabolite Changes after Local Cryotherapy in Knee Arthritis Patients. Metabolites. 2020 Nov 13;10(11):460. doi: 10.3390/metabo10110460. PMID 33202890
- [Result] De Boer AS, Van Lieshout EMM, Van Moolenbroek G, Verhofstad MHJ, Den Hartog D. Computer-Controlled Cooling in Operatively Treated Ankle or Hindfoot Fractures: A Retrospective Case-Control Study. J Foot Ankle Surg. 2021 Nov-Dec;60(6):1131-1136. doi: 10.1053/j.jfas.2021.04.014. Epub 2021 Apr 21. PMID 34039509
- [Result] Scheer RC, Newman JM, Zhou JJ, Oommen AJ, Naziri Q, Shah NV, Pascal SC, Penny GS, McKean JM, Tsai J, Uribe JA. Ankle Fracture Epidemiology in the United States: Patient-Related Trends and Mechanisms of Injury. J Foot Ankle Surg. 2020 May-Jun;59(3):479-483. doi: 10.1053/j.jfas.2019.09.016. PMID 32354504
- [Result] Lin S, Xie J, Yao X, Dai Z, Wu W. The Use of Cryotherapy for the Prevention of Wound Complications in the Treatment of Calcaneal Fractures. J Foot Ankle Surg. 2018 May-Jun;57(3):436-439. doi: 10.1053/j.jfas.2017.08.002. PMID 29685558
- [Result] Finger A, Teunis T, Hageman MG, Ziady ER, Ring D, Heng M. Association Between Opioid Intake and Disability After Surgical Management of Ankle Fractures. J Am Acad Orthop Surg. 2017 Jul;25(7):519-526. doi: 10.5435/JAAOS-D-16-00505. PMID 28574942

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT06396364/Prot_SAP_000.pdf